CLINICAL TRIAL: NCT05264571
Title: The ICCA Study (Early Identification of Candida in Intra-abdominal CAndidiasis)
Brief Title: Early Identification of Candida in Intra-abdominal Candidiasis
Acronym: ICCA
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: SYMCEL (Unknown)
Responsible Party: Principal Investigator, NOVY Emmanuel, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2021PI051
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Candida Sepsis; Candidiasis, Invasive; Peritonitis Infectious; Critically Ill
Keywords: intra abdominal candidiasis; candida; diagnostic method; metabolic profile; virulence
MeSH Terms: conditions — Candidiasis, Invasive; Critical Illness; Torulopsis | interventions — Metabolome; Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- critically ill adult patients with intra-abdominal infection: The ICCA study is an ancillary study of a non-interventional prospective cohort study (the pBDG2 study, NCT03997929) The pBDG 2 study has enrolled ICU patients with intra-abdominal infection requiring abdominal surgery. During the surgery, peritoneal fluid has been collected to identify the pathogens involved and guide anti-infective therapies. After the routine analyses, the remained peritoneal fluid was stored to create a biological collection.
  This biological collection, in which the content of bacterias and yeasts is known, will be analysed with the calscreener.
  Interventions: Diagnostic Test: calscreener; Other: Metabolic profile; Other: optical microscopy; Other: RTqPCR

INTERVENTIONS:
Diagnostic Test: calscreener — The calscreener (SYMCEL®) is a new diagnostic tool to rapidly identify the presence of pathogens in biological samples based on micrometabolic activity detection. All living cells produce heat by the chemical and physical processes of life; by monitoring the heat flow over time (J/s, W) a significant amount of information can be obtained regarding the biological system.
Other: Metabolic profile — The cal screener allows the measure of metabolic activity of pathogens directly from a sample (here, the peritoneal fluid).
  The heat production will be compared between peritoneal fluid, with or without addition of bacteria
Other: optical microscopy — To explain the metabolic activity, growth and yeast-to-hyphae transition will be analysed using optical microscopy and conventional culture
Other: RTqPCR — To explain the metabolic activity, level of expression of 5 Candida albicans virulence genes (UME6, ALS3, SFL2, HWP1 and ECE1) will be address and compared between peritoneal fluid.

SUMMARY:
Intra-abdominal candidiasis remains the first origin of invasive candidiasis in critically ill patients with a mortality up to 60%. This high mortality is partly related to delay of anti-fungal treatment administration. According to experts in the field, new diagnostic methods to rapidly detect Candida in intra-abdominal infections is mandatory because the current strategies suffer from a lack of both sensitivity and specificity.

The calscreener (SYMCEL®) is a new diagnostic tool to rapidly identify the presence of pathogens in biological samples based on micrometabolic activity detection. This technology also allows to measure the metabolic activity of pathogens.

The ICCA project will test the feasibility, the accuracy and the diagnostic performance of the calscreener on an existing biological collection of peritoneal fluid. This collection came from a cohort of critically ill patients with intra-abdominal infection which required abdominal surgery. Intra-abdominal infections consist of bacterial peritonitis and intra-abdominal candidiasis. The presence of pathogens (bacteria and yeast) is already known, the peritoneal fluid being stored after routine analysis (bacteriology / mycology).

In addition to the detection / identification of yeast will be investigated in this project, the cal screener will be used to evaluate the metabolic profile of Candida albicans in the peritoneal fluid, alone and with bacteria. This objective aims to evaluate the virulence of Candida in the peritoneal fluid from a metabolic perspective. The results will be compared to phenotypic and molecular evaluation.

DETAILED DESCRIPTION:
The high mortality rate of patients with intra-abdominal candidiasis infection is partly related to delay in anti-fungal treatment. The gold standard method for Candida detection remains the yeast culture on mycological media which suffers from a delayed response time (up to 5 days).

Consequently, in the routine practice, the decision to start an anti-fungal treatment is based on predictive scores such as the Peritonitis score. Whatever the score, they all suffer from a lack of sensitivity and specificity and could expose ICU patients to delayed treatment with negative impact on mortality. Once introduced and before the availability of the result of the culture, the anti-fungal can be stopped based on two serum measures of 1,3 beta D Glucan < 80 pg/ml. This strategy allows anti-fungal spare. Therefore, there is a room for improvement regarding early Candida detection and identification for the right choice of anti-fungal.

The calscreener (SYMCEL®) is a new diagnostic tool to rapidly identify the presence of pathogens in biological samples based on micrometabolic activity detection. The metabolic activity anticipates the future positive culture. To date, most of the experiments with the calscreenerTM concern bacteria. During the development phase, some experiments have been performed with Candida, mostly in vitro. Data of feasibility with clinical samples such as the peritoneal fluid are lacking. Besides, there is currently no library regarding the metabolic profile of Candida, in both albicans and non-albicans species. All in all, its routine use is currently impossible.

First results (unpublished data from our team) of metabolic activity detection in peritoneal fluid with known presence of Candida showed a time detection <1 hour. We aim to confirm these promising results using biological samples collected in an ongoing cohort study. We first need to describe the metabolic activity curves of different Candida species in order to constitute a library.

The heat production of each peritoneal fluid will be measured, and then compared considering the presence or absence of bacteria. Then, to explain the metabolic activity, a phenotypic evaluation of candida (growth and yeast-to-hyphae transition) and molecular evaluation (level of expression of virulence gene) will be performed.

ELIGIBILITY:
The criteria belong to the pBDG2 study (Peritoneal 1.3-ß-D-glucan for the Diagnosis of Intra-abdominal Candidiasis in Critically Ill Patients).

Inclusion Criteria:

* adult
* Covered by health insurance
* Admitted in ICU with intra-abdominal infection requiring abdominal surgery or percutaneous drainage

Exclusion Criteria:

* Pregnant or lactating woman
* Patient deprived of liberty after administration of juridical decision
* Patient under psychiatric care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the present study will be used the clinical samples issued from the biological collection of peritoneal fluid issue from the pBDG2 study. The presence of Candida of each sample is known thanks to routine analysis. According to the ethic committee, only peritoneal fluid issued from patients from the centre "NANCY" will be investigated in the ICCA STUDY.
  The results obtained with the calscreener will be compared to those obtain by yeast culture to confirm the Candida detection irrespective and depending on the albicans and non-albicans species.
  Lastly the delay of detection with the calscreener will be compared to the growth delay of yeast culture
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Detection (Yes/No) of the presence of Candida in the peritoneal fluid | Day 1 - 3
  Detection by the calscreener : detection of metabolic activity > 5 µW (according to SYMCEL recommendation)

SECONDARY OUTCOMES:
Delay (in hours) of detection | Day 1 - 3
  Delay (in hours) from the start of calscreener analysis to first detection of heat flow > 5 µW

OTHER OUTCOMES:
Heat production (Joule) | Day 1 - 3
  Heat production depending on the peritoneal fluid and the presence or absence of bacteria
Candida morphology | Day 1
  C. albicans SC5314 strain will be inoculated in triplicate into one mL of the different peritoneal fluid, as well as control media (Sabouraud and ascitic fluid) at an optical density (OD) of 0.3 nm, corresponding to approximately 3.10^6 colonies of C. albicans per millilitre (C. albicans/mL) of media. Control wells containing only the media without C. albicans were also included on the same 24-well plate to confirm the absence of contamination.
  The 24-well plate will be inoculated and incubated at 37°C with shaking at 300 RPM for 24 hours.
  The morphology of C. albicans (yeast or pseudo-hyphae or hyphae) was observed under a light microscope at hourly intervals for the initial eight hours, followed by observations at H16 and H24.
Candida growth | Day 1
  C. albicans SC5314 strain will be inoculated in triplicate into one mL of the different peritoneal fluid, as well as control media (Sabouraud and ascitic fluid) at an optical density (OD) of 0.3 nm, corresponding to approximately 3.10^6 colonies of C. albicans per millilitre (C. albicans/mL) of media. Control wells containing only the media without C. albicans were also included on the same 24-well plate to confirm the absence of contamination.
  The 24-well plate will be inoculated and incubated at 37°C with shaking at 300 RPM for 24 hours.
  C. albicans growth was assessed by inoculating 10 μL from each well onto SBD dextrose agar, and the colonies were counted after 24 hours of incubation at 37°C. To facilitate counting, 1000-fold dilutions of each inoculated well were prepared beforehand.
Candida virulence gene expression | Day 1
  C. albicans inoculation in the different media followed the same protocol as for phenotypic evaluation, with an overnight culture of 24h before gene expression analysis. The five virulence genes of interest are UME6, ALS3, SFL2, HWP1 and ECE1. After the 24-hour overnight culture, the samples will be centrifuged to retain only the cell pellet. The cell pellet was then washed twice with 10 mL of phosphate-buffered saline (PBS). Subsequently, the PBS was removed, leaving behind only the cell pellet. RNA extraction will be performed using the FASTPREP® lysis technology. Reverse transcription will be performed using the QuantiTect Reverse Transcription kit from Qiagen® (Germantown, Maryland, United States) following the manufacturer's instructions. The qPCR was performed in MicroAmp Optical 96-Well Reaction Plates (Applied Biosystems) using the CFX96 Real-Time PCR System (Bio-Rad, Marnes-la Coquette, France).

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novy E, Esposito M, Birckener J, Germain A, Losser MR, Machouart MC, Guerci P. Reappraisal of intra-abdominal candidiasis: insights from peritoneal fluid analysis. Intensive Care Med Exp. 2023 Sep 30;11(1):67. doi: 10.1186/s40635-023-00552-0. PMID 37776390